CLINICAL TRIAL: NCT00190788
Title: A Phase IIIb Study to Determine Efficacy and Safety of Extended Drotrecogin Alfa (Activated) Therapy in Patients With Persistent Requirement for Vasopressor Support After 96 Hour Infusion With Commercial Drotrecogin Alfa (Activated)
Brief Title: Extended Therapy of Drotrecogin Alfa (Activated) 4 vs 7 Days Infusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6001; F1K-MC-EVBQ
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Sepsis; Hypotension
MeSH Terms: conditions — Sepsis; Hypotension | interventions — drotrecogin alfa activated

INTERVENTIONS:
Drug: Drotrecogin Alfa (Activated)
Drug: placebo

SUMMARY:
The purpose of this study is to determine whether continued administration of Drotrecogin Alfa (Activated) up to additional 72 hours - after the so far recommended 96 hour infusion period - results in a more rapid resolution of hypotension in severe septic patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis patients treated with 96 hour infusion of commercial Drotrecogin Alfa (Activated)
* Continue requirement of Vasopressor support after 96 hour commercial infusion

Exclusion Criteria:

* Patients require extensive surgical procedures within next 3 days
* Patients with platelet count below 30,000/mm3
* Patients receiving therapeutic heparin of 15,000 units/day and more
* Patients not expected to survive 24 days
* Patients contraindicated as to the country specific registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
- To assess whether continued administration of Drotrecogin Alfa (Activated)for up to 72 additional hours after 96 hours infusion of commercial DDA results in more rapid resolution of vasopressor-dependent hypotension

SECONDARY OUTCOMES:
Evaluate Reduction of 28-day all cause mortality
Evaluate effects on various organ functions over 14 days
Evaluate effects on the concentration of various biomarkers
Investigate safety profile of an extended infusion of DDA

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Loma Linda, California, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris, France

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com